CLINICAL TRIAL: NCT06643585
Title: SURVIVE HERoes - A Randomized Secondary Adjuvant Treatment Intervention Study Comparing Trastuzumab-Deruxtecan to SOC Therapy in eBC Patients With Molecular Relapse
Brief Title: A Randomized Secondary Adjuvant Treatment Intervention Study Comparing Trastuzumab-Deruxtecan to SOC Therapy in eBC Patients With Molecular Relapse
Acronym: SURVIVE HERoes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Wolfgang Janni (Other)
Responsible Party: Sponsor-Investigator, Prof. Wolfgang Janni, Prof. Dr. med. Wolfgang Janni, University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURVIVE HERoes; 2024-516173-76-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Trastuzumab-Deruxtecan (i.v. 5,4 mg/kg, q3w) + endocrine therapy (if hormonal-receptor-positive) for 16 cycles or until relapse, if earlier
  Interventions: Drug: Trastuzumab-Deruxtecan
- Arm B (Active Comparator): Continuous treatment of physician's choice (may include endocrine treatment, CDK4/6-Inhibition, T-DM1, Olaparib, Trastuzumab, Pertuzumab, Capecitabine or Neratinib)
  Interventions: Other: Physicians Choice (PhC).

INTERVENTIONS:
Drug: Trastuzumab-Deruxtecan — Trastuzumab-Deruxtecan (i.v. 5,4 mg/kg, q3w) + endocrine therapy (if hormonal-receptor-positive) for 16 cycles or until relapse, if earlier
  Arms: Arm A
Other: Physicians Choice (PhC). — Continuous treatment of physician's choice (may include endocrine treatment, CDK4/6-Inhibition, T-DM1, Olaparib, Trastuzumab, Pertuzumab, Capecitabine or Neratinib)
  Arms: Arm B

SUMMARY:
Prospective, multi-center, randomized, open label comparative Phase III study in patients with intermediate to high-risk (as defined in the SURVIVE trial) HER2-positive or HER2-low early breast cancer, who participate in the SURVIVE trial and experience a molecular relapse, as assessed based on a positive circulating tumor DNA (ctDNA) result, with 2:1 allocation to:

* Arm A: Trastuzumab-Deruxtecan (i.v. 5,4 mg/kg, q3w) + endocrine therapy (if hormonal-receptor-positive) for 16 cycles or until relapse, if earlier
* Arm B: Continuous treatment of physician's choice (may include endocrine treatment, CDK4/6-Inhibition, T-DM1, Olaparib, Trastuzumab, Pertuzumab, Capecitabine or Neratinib)

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for study participation if they comply with the following criteria:

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Females or males, ≥ 18 years and ≤ 75 years of age.
3. Invasive breast carcinoma as revealed by local pathology that is either:

   1. HER2-positive defined as an immunohistochemistry (IHC) score of 3+ and/or positive by in situ hybridization (ISH) in Her2 2+ tumors (as defined in 2018 American Society of Clinical Oncology - College of American Pathologists [ASCO-CAP] guidelines)
   2. HER2-low defined as an immunohistochemistry (IHC) score of 1+ or an IHC score of 2+ with a mandatory negative in situ hybridization (ISH), as defined in 2018 American Society of Clinical Oncology - College of American Pathologists [ASCO-CAP] guidelines.
4. Complete resection of the tumor with resection margins free of invasive carcinoma (R0).
5. Participation in the SURVIVE study and evidence of molecular relapse (as assessed based on a positive ctDNA result obtained in the SURVIVE-study)
6. No evidence of metastatic relapse as revealed by a CT-scan (Abdomen/Chest) and a SPECT bone scan that must be performed within 8 weeks before randomization (M0).
7. Completion of surgery, (neo-)adjuvant chemotherapy (if applicable) and radiation therapy (if applicable, whichever occurred last) at least 6 months before randomization.
8. Adjuvant/Postneoadjuvant treatment with Trastuzumab, Pertuzumab, T-DM1, Capecitabine, Pembrolizumab, and Olaparib must be discontinued upon randomization into Arm A (treatment with trastuzumab deruxtecan). The washout periods (see Table 2) must be complied with. Endocrine therapy (i.e. Tamoxifen, Letrozol, Anastrozol, Fulvestrant or Exemestane) can be administered simultaneously to treatment with trastuzumab deruxtecan.
9. Known HR status, per local laboratory assessment, as defined by ASCO-CAP guidelines (≥1%): HR-positive status defined by either positive estrogen receptor (ER) and/or positive progesterone receptor (PR) status. HR-negative status defined by both known negative ER and known negative PR
10. Left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to randomization
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at Screening
12. Adequate organ and bone marrow function within 28 days before randomization as described in table 1. Organ and bone marrow function criteria must also be met when laboratory tests are repeated within 3 days before Cycle 1 Day 1. Transfusion (red blood cell or platelet) or G-CSF administration is not allowed within 2 weeks prior to the day on which marrow function is assessed.
13. Adequate treatment washout period before treatment with trastuzumab deruxtecan (in case of randomization into cohort A), defined in table 2.
14. Female subjects: Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of Investigational Medicinal Product (IMP).

    1. Women of childbearing potential are defined as those who are not surgically sterile (underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause.
    2. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception (see 5.5.1.) from the time of screening and must agree to continue using such precautions for 7 months after the last dose of IMP. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
    3. Female subjects must not donate, or retrieve for their own use, ova from the time of randomization and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.
15. Male subjects: Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period, as described in section 5.5.1. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of randomization/enrolment, throughout the study and for 4 months after the last dose of IMP. Preservation of sperm should be considered prior to enrolment in this study.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer.
2. Patients with a history of any secondary primary malignancy are ineligible with the following exceptions:

   * ipsi- or contralateral non-invasive carcinoma of the breast (DCIS)
   * other, curatively treated in-situ disease
   * adequately treated non-melanoma carcinoma of the skin
3. Prior treatment with T-DXd.
4. Combination of T-DXd with any other anti-cancer treatment is not permitted, except for endocrine therapy.
5. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
6. Patients with a medical history of myocardial infarction (MI) within 6 months before first exposure to study intervention, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI.
7. Corrected QT interval (QTcF) prolongation to > 470 msec (females) or > 450 msec (males) based on average of the screening triplicate 12-lead ECG.
8. History of (non-infectious) Interstitial lung disease (ILD) / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
9. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
10. Active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects should be tested for HIV prior to randomization/enrolment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
11. Lung criteria:

    1. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (for example pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
    2. Any autoimmune, connective tissue or inflammatory disorders (for example Rheumatoid arthritis, Sjogren's, sarcoidosis et cetera) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the electronic case report form (eCRF) for patients who are included in the study.
    3. Prior pneumonectomy (complete)
12. Participants with past or resolved HBV infection are eligible only if they meet all of the following criteria:

    * HBsAg (-) (for > 6 months off anti-viral treatment),
    * Anti-HBc (+) (IgG or total Ig),
    * HBV DNA undetectable,
    * Liver architecture normal (absence of any liver pathology including absence of cirrhosis or fibrosis on prior imaging or biopsy,
    * Absence of HCV co-infection or history of HCV co-infection.
    * Access to a local Hepatitis B expert during and after the study. Such participants should be closely monitored for HBV reactivation.
13. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of T-DXd.

    Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP.
14. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline.

    Note: Toxicities related to endocrine therapy should be documented but does not lead to exclusion of patient from the study.

    Also, subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to first exposure to study intervention and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as:
    1. Chemotherapy-induced neuropathy
    2. Fatigue
    3. Residual toxicities from prior immune-oncology treatment: Grade 1 or Grade 2 endocrinopathies which may include:

    i. Hypothyroidism/hyperthyroidism ii. Type 1 diabetes iii. Hyperglycemia iv. Adrenal insufficiency v. Adrenalitis vi. Skin hypopigmentation (vitiligo)
15. Known allergy or hypersensitivity to study treatment or any of the study drug excipients.
16. History of severe hypersensitivity reactions to other monoclonal antibodies.
17. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2032-04-22 (Estimated); Study Completion 2032-04-22 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance rate 12 months after randomization | from enrollment to end of treatment after 12 months
  To compare ctDNA clearance rate twelve months after randomization between patients in the experimental arm (Arm A) versus patients in the standard of care arm (Arm B). ctDNA is measured as per RaDaR assay (see 5.8).
  Endpoint:
  ctDNA clearance rate is defined as the proportion of patients with a ctDNA negative blood test result at a given time point: (Patients with negative cfDNA at 12 months)/(all patients)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Ulm, Ulm, Germany